CLINICAL TRIAL: NCT06646978
Title: Long-term Risk of Second Primary Malignancies for Chronic Myeloid Leukaemia in the French Imatinib-based SPIRIT Trial
Acronym: K2SPIRIT
Status: Enrolling by invitation | Type: Observational
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2SPIRIT
Record Dates: First submitted 2024-10-14; First posted 2024-10-17 (Actual); Last update posted 2024-10-17 (Actual); Status verified 2024-10

CONDITIONS: Chronic Myeloid Leukemia (CML)
Keywords: second primary malignancies; imatinib
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — Imatinib Mesylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients with chronic myeloid leukaemia included in the French imatinib-based SPIRIT trial
  Interventions: Drug: Imatinib (STI571)

INTERVENTIONS:
Drug: Imatinib (STI571) — Imatinib-based regimen

SUMMARY:
Imatinib is a tyrosine kinase inhibitor that has improved the prognosis of patients with chronic myeloid leukemia (CML). CML has become a chronic disease requiring long-term administration of imatinib. Late adverse effects were initially unknown. Since 2005, imatinib has been suspected to increase the risk of second primary malignancies (SPM). Through the French "STI571 Prospective Randomized Trial" (SPIRIT), we studied the incidence of SPM after more than 20 years of exposure, and treatment strategies for CML and SPM at their occurrence.

ELIGIBILITY:
Inclusion Criteria:

* Included in the French SPIRIT trial

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with chronic myeloid leukaemia included in the French imatinib-based SPIRIT trial
Sampling Method: Non-Probability Sample
Enrollment: 787 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Risk of second primary malignancies (SPM) | Through study completion, an average of 20 years
  SPM is an invasive primary cancer diagnosed at least 6 months after CML diagnosis. Non-melanoma skin cancers were excluded from the analysis.

SECONDARY OUTCOMES:
Treatment strategies for CML and SPM at their occurrence | At the occurence of SPM. Through study completion, on average 20 years
  For treatment strategy of CML: response, modification of treatment (temporary discontinuation, permanent interruption, replace by a new generation TKI), relapse.
  For treatment strategy of SPM: intent of treatment (curative, palliative, follow without treatment), type of treatment (surgery, radiotherapy, chemotherapy, targeted therapy), atypical adverses events, modification of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Preudhomme C, Guilhot J, Nicolini FE, Guerci-Bresler A, Rigal-Huguet F, Maloisel F, Coiteux V, Gardembas M, Berthou C, Vekhoff A, Rea D, Jourdan E, Allard C, Delmer A, Rousselot P, Legros L, Berger M, Corm S, Etienne G, Roche-Lestienne C, Eclache V, Mahon FX, Guilhot F; SPIRIT Investigators; France Intergroupe des Leucemies Myeloides Chroniques (Fi-LMC). Imatinib plus peginterferon alfa-2a in chronic myeloid leukemia. N Engl J Med. 2010 Dec 23;363(26):2511-21. doi: 10.1056/NEJMoa1004095. PMID 21175313